CLINICAL TRIAL: NCT02695940
Title: A Phase 2a, Proof of Concept Trial, Testing Twice Daily Application of LEO 124249 Ointment 30 mg/g in the Treatment of Mild to Moderate Inverse Psoriasis
Brief Title: Trial Twice Daily Application of LEO 124249 Ointment 30 mg/g in Treatment of Mild to Moderate Inverse Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0133-1182
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Inverse Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 124249 ointment 30 mg/g (Active Comparator): Drug LEO 124249 ointment 30 mg/g twice daily application for 6 weeks, maximum of 1.44 g ointment per day
  Interventions: Drug: LEO 124249 ointment 30 mg/g
- LEO 124249 ointment vehicle (Placebo Comparator): LEO 124249 ointment vehicle twice daily application for 6 weeks, maximum of 1.44 g ointment per day
  Interventions: Other: LEO 124249 ointment vehicle

INTERVENTIONS:
Drug: LEO 124249 ointment 30 mg/g
  Arms: LEO 124249 ointment 30 mg/g
Other: LEO 124249 ointment vehicle
  Arms: LEO 124249 ointment vehicle

SUMMARY:
This is a phase 2a trial testing twice daily administration of LEO 124249 ointment 30 mg/g in the treatment of mild to moderate inverse psoriasis. Patients will be treated for 6 weeks, and the efficacy and safety will be compared with the treatment of LEO 124249 ointment vehicle.

DETAILED DESCRIPTION:
Single country, Multi-center, prospective, randomised, double-blind, 2 arms parallel-group, vehicle-controlled, 6 weeks, phase 2a trial in subjects with mild to moderate inverse psoriasis. LEO 124249 ointment 30 mg/g and LEO 124249 ointment vehicle treatments will be compared with regards to efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent prior to any trial specific procedures
* Male or female subjects between 18 to 75 years
* A diagnosis of stable mild to moderate inverse psoriasis (i.e. axillae, the infra- and intermammary, genital, scrotum, abdominal and retroauricular folds; the intergluteal cleft and perianal skin, in addition to neck or other skin folds). Mild to moderate is defined as having at least score 1 for each individual sign thickness and redness, and total TSS score of at least 5.
* The total treatment area can be up to 4% BSA (720 cm2).
* Subjects must have a history of psoriasis, or have psoriasis, or present with characteristic psoriasis leasons elsewhere on the body (including the scalp) at Visit 1 (Screening)
* Stable inverse psoriasis based on TSS evaluated at Visit 1 (Screening) and at Visit 2 (Start of treatment), which must not differ more than 1 point in any single clinical sign score (redness, scaling and thickness)
* Except for inverse psoriasis, overall good health including well controlled diseases (e.g. hypertension, diabetes, and thyroid disease) as determined by medical history, physical examination, electrocardiogram (ECG), vital signs (blood pressure, heart rate and body temperature) and clinical laboratory evaluation

Exclusion Criteria:

* Female subjects who are breastfeeding or pregnant
* Severe chronic inverse psoriasis, or psoriasis on the body (>30% of BSA)
* Current diagnosis of acute guttate, erythrodermic, exfoliative or pustular psoriasis
* Signs of viral (e.g. herpes or varicella) lesions of the skin, or signs of clinically active fungal or bacterial infection in any of the inverse psoriasis areas, as judged by the investigator
* Use of biological therapies (marketed/not marketed) with a possible effect on inverse psoriasis within 4 weeks (etanercept), 8 weeks (adalimumab, alefacept, infliximab), 16 weeks (ustekinumab, secukinumab) or 4 weeks/5 half-lives (whichever is longer) for experimental biological products prior to Visit 2 (Start of treatment)
* Use of systemic treatments (marketed/non-marketed), other than biologics, with a potential effect on inverse psoriasis (e.g., corticosteroids, retinoids, dimethylfumarate, cyclosporine, azathioprine methotrexate, immunosuppressants) within 6 weeks prior to Visit 2 (Start of treatment) (inhaled or intranasal steroids corresponding of up to 1 mg prednisone for asthma or rhinitis may be used)
* Use of very potent topical corticosteroids (WHO group IV) for the treatment of psoriasis on the body and/or scalp within 4 weeks prior to Visit 2 (Start of treatment)
* Use of topical medication for the treatment of inverse psoriasis: WHO group I-III corticosteroids, retinoids, vitamin D analogues, immunomodulators (e.g. macrolides, calcineurin), anthracen derivatives, tar, or salicylic acid within 2 weeks prior to Visit 2 (Start of treatment)
* Exposure to phototherapy (PUVA, UVA, UVB, Grenz Ray therapy) within 4 weeks prior to Visit 2 (Start of treatment)
* Subjects with a positive HBV score antibody, HBsAg, anti-HCV or anti-HIV test at Visit 1 (Screening)
* Subjects with history of an immunocompromising disease (e.g., lymphoma, HIV, Wiskott-Aldrich Syndrome)
* Any current dermatological disorder (e.g. serborrhic dermatitis, contact dermatitis, cutaneous mycosis) which may confound the evaluation of inverse psoriasis
* Known malignancy (other than cervical carcinoma in situ, basal cell or squamous cell carcinoma) within 5 years before Visit 1 (Screening)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The total sign score (TSS) at Week 6 (Visit 6) | after 6 weeks of treatment

SECONDARY OUTCOMES:
For PGA, the number of subjects reaching controlled disease at Visit 6 (Week 6) | after 6 weeks of treatment
Score for clinical sign redness for inverse psoriasis: (score 0 to 4) at Visit 6 (Week 6) | after 6 weeks of treatment
Score for clinical sign thickness for inverse psoriasis: (score 0 to 4) at Visit 6 (Week 6) | after 6 weeks of treatment
Score for clinical sign scaliness for inverse psoriasis: (score 0 to 4) at Visit 6 (Week 6) | after 6 weeks of treatment
Size of treatment area of inverse psoriasis at Visit 6 (Week 6) | after 6 weeks of treatment
For PaGA, the number of subjects reaching controlled disease at Visit 6 (Week 6) | after 6 weeks of treatment
Dermatology Life Quality Index (DLQI) questionnaire at Visit 6 (Week 6) | after 6 weeks of treatment
Treatment satisfaction questionnaire for medication (TSQM II) at Visit 6 (Week 6) | after 6 weeks of treatment
Subjects assessment of itching (daily assessment in diary of the first 14 days on treatment (between Visits 2 (Start of treatment) to 4 (Week 2), followed by assessments at the following Visits 4 (Week 2) to 6 (Week 6)) | after 6 weeks of treatment
Subjects overall assessment of cosmetic acceptability at Visit 6 (Week 6) | after 6 weeks of treatment
Evaluation of population steady state pharmacokinetics of LEO 124249 at Visit 3 (Week 1), by sampling of 1 blood sample to get 1 plasma concentration value per patient after 1 weeks treatment | after 6 weeks of treatment
Adverse Events | after 6 weeks of treatment
Abnormal and clinically significant findings in blood pressure, heart rate, body temperature will be listed | after 6 weeks of treatment
Abnormal and clinically significant laboratory parameters will be listed | after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Luger, MD, Principal Investigator — Universitätsklinikum Münster, Klinik fur Hautkrankheiten
Locations (1):
- Johannes Niesmann, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: LEO Pharma Clinical Trials — https://www.leopharmatrials.com/en